CLINICAL TRIAL: NCT06192667
Title: 24- Month Clinical Performance of Injectable and Conventional Resin Composites in Class I Cavities
Brief Title: Clinical Performance of Injectable Composite Resins in Class I Cavities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslı Ceren Terzi, Principal İnvestigator, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KA-22112
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Caries,Dental
Keywords: Conventional resin composite; Injectable resin composite; Class I restoration
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Geanial Injectable Composite Resin (Experimental): It contains 31% methacrylate monomer in the resin matrix and 69% silica and barium glass as fillers. A1, A2, A3, A3.5, A4, B1, B2, B3, C3, CV, BW, AO2, AO3, JE, AE colors are available. Due to their high durability, they can be used in places where recyclable composite resins are used. Apart from this, they are used as fissure sealants, sealants, repair of indirect restorations, blocking of undercuts and liner, like flowable composites.
  After completing the cavity, the enamel surface was selectively roughened using 37% orthophosphoric acid for 15 seconds. Subsequently, G2 Bond Universal adhesive agent (GC Corp., Tokyo, Japan) was utilized. It was applied in 2mm layers in accordance with the composite manufacturer's instructions. Each layer was polymerized for 20 seconds.
  Interventions: Device: GC Geanial Injectable (Tokyo,Japan)
- 3M Filtek Z250 Universal Restorative (Experimental): It is designed to be used in both anterior and posterior restorations. The filler in the Filtek Z250 restorative is zirconia/silica. The inorganic filler is 60 vol% (without silane treatment) with a particle size of 0.01 to 3.5 μm. Filtek Z250 restorative contains BIS-GMA, UDMA and BIS-EMA monomers. Various restorative color options are available. It is packaged in conventional syringes and single-dose capsules.
  After completing the cavity, the enamel surface was selectively roughened using 37% orthophosphoric acid for 15 seconds. Subsequently, G2 Bond Universal adhesive agent (GC Corp., Tokyo, Japan) was utilized. It was applied in 2mm layers in accordance with the composite manufacturer's instructions. Each layer was polymerized for 20 seconds.
  Interventions: Device: 3M Filtek Z250 Universal Restorative (Germany)

INTERVENTIONS:
Device: GC Geanial Injectable (Tokyo,Japan) — Highly filled composite resin
  Arms: Geanial Injectable Composite Resin
Device: 3M Filtek Z250 Universal Restorative (Germany) — Conventional composite resin
  Arms: 3M Filtek Z250 Universal Restorative

SUMMARY:
Purpose of research: Evaluation and comparison of 24-month clinical performance of injectable and conventional resin composites in class I cavities.

DETAILED DESCRIPTION:
The mechanical properties of conventional resin composites have been tried to be improved. In addition to the developed mechanical properties, the need for easy and fast application led to the development of flowable composites. Flowable composites have lower filler ratio than conventional hybrid composites so they are less rigid and have lower modulus of elasticity. For these reasons, the use of flowable composites in areas that may be exposed to high forces, especially occlusal cavities, is not recommended. Today, it is aimed to increase the wear resistance by increasing the amount of filler in flowable composites and producing injectable composites. A new product recently introduced to the market, a high-strength nano-filled injectable composite material, GC's G-ænial Universal Injectable(Tokyo,Japan), was also included in the study. This is a low-viscosity composite in which modifications have been made to provide a product with high wear resistance and depth of cure to make it suitable for posterior restorations.

One lesion in each patient will be randomly assigned to be restored using either the G-aenial Universal Injectable or Filtek Z250 resin composites. The adhesive, G2-BOND Universal will be used for adhesive procedures. The clinical procedure for the restorations will be performed by a single operator. The restorations will be evaluated by two calibrated examiners at baseline and at 6, 12, 18, 24 months in accordance with the modified USPHS criteria. Data will be statistically analyzed using the Chi-square and Cochran Q tests (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals who do not have any systemic disease that prevents restorative treatment
* Individuals between the ages of 18-35
* Brushing your teeth twice a day
* Having at least 20 teeth in occlusion and at least 2 occlusal lesions with antagonist teeth in the opposite arch
* Volunteer individuals who agree to participate in the research and sign the informed consent form and who have undergone initial periodontal treatment will be included in the study.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Individuals with advanced periodontal disease
* Individuals using removable partial dentures
* Individuals with bruxism
* Individuals with malocclusion
* Patients with known allergies to resin-based restorative materials and bonding agents
* Patients with a history of allergy to local anesthesia
* Endodontic treatment, teeth that need pulp capping or endodontic treatment is available

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Marginal Adaptation | From baseline to 24 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding marginal adaptation. Marginal adaptation was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed . Scores; Alfa: Closely adapted, no visible crevice. Bravo: Visible crevice, explorer will penetrate. Charlie: Crevice in which dentin is exposed
Marginal Staining | From baseline to 24 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding marginal staining. Marginal staining was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed . Scores: Alfa: No discoloration. Bravo: Discoloration without. Charlie: Discoloration with penetration in pulpal direction
Retention | From baseline to 24 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding retention rate. Retention rate was evaluated by 2 independent clinicians. Scores: Alfa: No loss of restorative material. Charlie: Any loss of restorative material
Postoperative sensitivity | From baseline to 24 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding retention rate. Retention rate was evaluated by 2 independent clinicians. Scores: Alfa: Not present. Bravo: sensitive but diminishing in intensity. Charlie:constant sensitivity, not diminishing in intensity
Seconder caries | From baseline to 24 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding retention rate. Retention rate was evaluated by 2 independent clinicians. Scores: Alfa: No caries present. Charlie: Caries present

CONTACTS AND LOCATIONS:
Overall Officials: Cansu Atalay, Assoc. Prof., Principal Investigator — Hacettepe University; Aslı Ceren Terzi, Principal Investigator — Hacettepe University; Esra Ergin, Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shaalan OO, Abou-Auf E. A 24-Month Evaluation of Self-Adhering Flowable Composite Compared to Conventional Flowable Composite in Conservative Simple Occlusal Restorations: A Randomized Clinical Trial. Contemp Clin Dent. 2021 Oct-Dec;12(4):368-375. doi: 10.4103/ccd.ccd_600_20. Epub 2021 Dec 21. PMID 35068835
- [Background] Ypei Gia NR, Sampaio CS, Higashi C, Sakamoto A Jr, Hirata R. The injectable resin composite restorative technique: A case report. J Esthet Restor Dent. 2021 Apr;33(3):404-414. doi: 10.1111/jerd.12650. Epub 2020 Sep 11. PMID 32918395
- See also: Related Info — https://europe.gc.dental/tr-TR/products/gaenialuniversalinjectable